CLINICAL TRIAL: NCT00462904
Title: Phase IIa Trial to Evaluate the Pharmacokinetic Response to Bactericidal/Permeability-increasing Protein (rBPI21) for the Treatment of Patients With Burn Injury.
Brief Title: Pharmacokinetic Response to BPI in Burns
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Xoma to no longer supply drug for the study
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Joseph P. Minei, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XO-400761
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BPI infusion group (Experimental): BPI will be infused by bolus for 30 minutes followed by continuous infusion for 47.5 hours
  Interventions: Drug: BPI

INTERVENTIONS:
Drug: BPI — BPI will be give IV with an initial bolus given over 30 minutes and then a continuous infusion for the next 47.5 hours
  Other Names: Opebacan

SUMMARY:
The purpose of this study is to evaluate the safety of a protein called BPI that is naturally made by the body's white blood cells to fight infection.

DETAILED DESCRIPTION:
This study will initially evaluate an FDA approved investigational dosage and will measure the blood levels over time while BPI is being infused through a vein to see if the dose is potentially enough to obtain the desired effect. The drug will be started within 8 hours of burn injury and continued for 48 hours. Patients will be followed on admission and through infusion in the Burn ICU where they will be monitored by ICU standards. They will be seen regularly thereafter on post-burn days 1, 2, 3, 4, 7, 14 and 28 days while in the hospital. If the patient is discharged prior to the 28 day evaluation, they will be evaluated on or around the 28th day in the burn clinic. A blood sample will be obtained to look for potential genetic markers that may increase a burn patients' risk to develop infection in the post burn period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13 years to 60 years old
* Sustained partial-thickness or full-thickness burn greater than 20% and less than 41% TBSA
* Parental consent (if subject is less than 18 years old) or individual (if subject is equal to or older than 18) signed, informed consent.
* Able to start BPI in infusion within 8 hours of burn injury.

Exclusion Criteria:

* Age > 61.
* Inhalational injury requiring mechanical ventilation.
* Partial and full thickness burns totaling > 41% total body surface area
* Cardiac dysfunction, defined as the presence of any of the following:

  1. New York Heart Class 3 or 4 heart failure.
  2. Unstable angina or acute myocardial infarction.
  3. Left ventricular ejection fraction known to be < 35%.
* Electrical or lightening induced burn injury or any injury that required cardio-pulmonary resuscitation.
* Concomitant non-burn trauma with an ISS > 9.
* Non-survivable injury secondary to burn size - patients made DNR or comfort care due to burn size.
* Patients with known causes of immunosuppression:

  1. Known history of HIV/AIDS
  2. Chronic steroid use for underlying medical conditions (equivalent to 15 mg prednisone/day).
  3. Active oncolytic therapy for known malignancy
* Known or suspected pregnancy
* Known allergy to rBPI21

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Minei, MD, Principal Investigator — UT Southwesten Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BPI Infusion Group
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | BPI Infusion Group
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Plasma Levels of BPI
Description: pharmacokinetic data over the 48 hour infusion period will be obtained as well as 24 hours post infusion.
Time Frame: 48 hours of infusion and 24 hours post infusion
Population: This study was terminated early by the sponsor. Ownership of the company changed, and there was no longer a desire to continue the trial; therefore, no analysis was performed. No data was collected.
Arm/Group | BPI Infusion Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety Parameters
Description: Routine physiologic and laboratory parameters will be followed for 28 days post infusion. These will include vital signs, cardiac enzymes, renal and hepatic function.
Time Frame: 28 days
Population: as for outcome 1
Arm/Group | BPI Infusion Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: study suspended
Arm/Group | BPI Infusion Group
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPI Infusion Group (N=4)
PAIN (Pregnancy, puerperium and perinatal conditions) | 1 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPI Infusion Group (N=4)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
ACIDOSIS (Metabolism and nutrition disorders) | 2 (2)
AGGITATION (Psychiatric disorders) | 1 (1)
ALKALOSIS (Metabolism and nutrition disorders) | 1 (5)
ANEMIA (Blood and lymphatic system disorders) | 4 (5)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
AZOTEMIA (Renal and urinary disorders) | 3 (5)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CELLULITIS/ABSCESS (Infections and infestations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DECREASED PRE-ALBUMIN (Investigations) | 2 (2)
FEVER (General disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 1 (1)
HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HYPERCHLORIDEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Ileus, GI (Gastrointestinal disorders) | 1 (1)
Increased C-Reactive Protein (Investigations) | 1 (1)
Increased CRP (Investigations) | 1 (1)
Infection Bladder (Infections and infestations) | 1 (1)
Infection Pneumonia (Infections and infestations) | 1 (1)
Infection Cellulitis (Infections and infestations) | 1 (1)
Infection Skin (Infections and infestations) | 1 (1)
Infection Skin Cellulitis (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (3)
Oversedation (Injury, poisoning and procedural complications) | 1 (1)
Pain (Investigations) | 1 (1)
Polycythemia (Blood and lymphatic system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 4 (4)
Vol Overload (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No